CLINICAL TRIAL: NCT03082404
Title: Effects of High-intensity Inspiratory Muscle Training in Chronic Kidney Disease: Randomized Clinical Trial
Brief Title: Inspiratory Muscle Training in Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Principal Investigator, Rodrigo Della Méa Plentz, PhD, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIIMT_CKD
Record Dates: First submitted 2017-03-12; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease; Inspiratory muscle training
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training group (Experimental): Six times a week (three supervised at hemodialysis unit and other three times at home), 5 series, 10 repetitions, two-minutes interval or according to the patient tolerance.
  Interventions: Other: Inspiratory muscle training
- Control group (No Intervention): The patients in this group will be evaluated at baseline and reassessed after five weeks of follow-up.

INTERVENTIONS:
Other: Inspiratory muscle training — Inspiratory muscle training will be performed during the first hour of hemodialysis treatment and the protocol will consist of five series with 10 repetitions, each series with a two-minute interval of according to patient tolerance. The overload will be adjusted weekly, beginning with 50% of the maximum inspiratory pressure, during the first week, 60% of maximum inspiratory pressure in the second and third week and 70% of maximum inspiratory pressure in the fourth and fifth weeks. Maximum inspiratory pressure will be evaluated before the protocol period and adjusted weekly by manovacuometry.
  Other Names: High intensity inspiratory muscle training
  Arms: Inspiratory muscle training group

SUMMARY:
Chronic kidney disease is a renal injury and progressive and irreversible loss of kidney function and in its most advanced stage is called chronic renal failure. Although hemodialysis replace some kidney function, patients suffer some alterations characterized by "uremic syndrome" typically expressed by: motor neuropathy and/ or autonomic neuropathy, cardiac or musculoskeletal myopathies, peripheral vascular changes, among others. Thereby, the the adoption of physical exercise should be encouraged. However, it is known that the ability to exercise the subject in hemodialysis is low and they present weakness of the peripheral muscular system, including inspiratory muscles. The aim of this study is to assess the effects of inspiratory muscle training (IMT) on ventilatory muscle strength and functional capacity of patients with chronic kidney disease in hemodialysis. For this the following assessments will be performed before and after intervention: six-minute walk test to functional capacity; Kidney Disease and Quality of Life - Short Form questionnaire for quality of life; flow-mediated dilatation to endothelial function; sit-to-stand test for proximal strength of lower limbs. The subjects will be randomized into two groups, IMTG (inspiratory muscle training group) and CG (control group). The first will receive the IMT, for five weeks, three times a week, during hemodialysis session and the patients will be oriented to realize more three days at home. The control group only will be evaluated and re-evaluated. Expected results at the end of the protocol with IMT are: increased inspiratory muscle strength; longest distance covered on the six-minute walk test; improved quality of life; increased muscle strength of the lower limbs; improved endothelial function.

DETAILED DESCRIPTION:
The research will be developed in the hemodialysis unit of the Santa Clara hospital of Santa Casa de Misericórdia de Porto Alegre. After the selection of patients for eligibility criteria they will be randomized into IMTG or control group. First all patients will be evaluated, and subsequently the patients in the IMTG will be trained six times per week (three times at hemodialysis unit and three times at home) for five weeks using a linear pressure load device (POWERbreathe Plus Light Resistance@, England). The sessions will take place in the first hour of dialysis and the training protocol will consist of five series with 10 repetitions, each serie with a two-minute interval or according to the patient´s feedback, using the Borg modified scale. The overload will be adjusted weekly, beginning with 50% of maximum inspiratory pressure and increasing until 70% along the protocol period. At the end of follow-up, both groups will be evaluated in order to compare.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease on hemodialysis for more than 3 months;
* Clearance of urea during hemodialysis (Kt/V ≥ 1.2).

Exclusion Criteria:

* Cognitive impairment that prevents conducting evaluations, as well as inability to understand and sign the informed consent form;
* Patients with recent sequel of stroke;
* Disabling musculoskeletal disease;
* Uncontrolled hypertension (Systolic blood pressure > 230 mmHg and diastolic blood pressure > 120 mmHg);
* Grade IV heart failure (NYHA) or decompensated;
* Uncontrolled diabetes (blood glucose > 300 mg/dL);
* Unstable angina;
* Fever and/or infectious disease;
* Recent acute myocardial infarction (two months);
* Active smokers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-04-03 (Estimated); Primary Completion 2017-05-02 (Estimated); Study Completion 2017-06-02 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | Five weeks
  Functional capacity will be assessed by the distance walked in six-minute walk test (6MWT)

SECONDARY OUTCOMES:
Muscle strength of inspiratory muscle | Five weeks
  Muscle strength will be assessed by manovacuometry
Proximal strength of lower limbs | Five weeks
  Proximal strength of lower limbs will be assessed by the number of repetitions performed in sit-and-stand test (SST).
Endothelial function | Five weeks
  Endothelial function will be assessed by flow mediated dilation technique
Quality of Life | Five weeks
  The quality of life will be assessed by questionnaire Kidney Disease and Quality-of-Life Short-Form (KDQOL-SFTM)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo DM Plentz, PhD, Principal Investigator — Federal University of Health Sciences of Porto Alegre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dipp T, Macagnan FE, Schardong J, Fernandes RO, Lemos LC, Plentz RDM. Short period of high-intensity inspiratory muscle training improves inspiratory muscle strength in patients with chronic kidney disease on hemodialysis: a randomized controlled trial. Braz J Phys Ther. 2020 May-Jun;24(3):280-286. doi: 10.1016/j.bjpt.2019.04.003. Epub 2019 May 6. PMID 31122717